CLINICAL TRIAL: NCT00332085
Title: Pilot Trial of Chromium-Metformin Combination in Type 2 Diabetes: Impact on Blood Sugar Control and Insulin Resistance
Brief Title: Pilot Trial of Chromium-Metformin Combination in Type 2 Diabetes
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Issues w/recruitment
Sponsor: Bastyr University (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 190
Record Dates: First submitted 2006-05-30; First posted 2006-06-01 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — picolinic acid

INTERVENTIONS:
Drug: Chromium Picolinate

SUMMARY:
This pilot trial seeks to gather preliminary data on the combination of chromium picolinate, the most commonly used form of chromium, and metformin. The trial will recruit type 2 diabetes subjects already on metformin and treat them with chromium for 8 weeks. The results of this trial will provide vital preliminary data including safety and size of effect to direct future studies.

DETAILED DESCRIPTION:
Chromium is widely marketed for use in diabetes and is used as a dietary supplement by approximately 10 million US consumers, second only to calcium supplementation. Limited scientific research has supported the potential of chromium to be beneficial in diabetes to improve blood sugar control and insulin sensitivity, yet many of these studies have design flaws and the relevance of the research in the US population has been questioned. Research on use of complementary & alternative medicine (CAM) suggests as many as 40% use CAM in combination with conventional medicine. Research performed at the Bastyr Center for Natural Health suggests 69% of patients get chromium as part of their treatment and 45% are on oral medications for blood sugar control. Metformin is the most commonly prescribed oral medication for diabetes in the world. The combination of chromium and metformin has never been studied in a clinical trial despite frequent use in combination. Additionally, research suggests chromium and metformin share at least one mechanism of action leading to questions about possible interactions - both favorable and unfavorable - resulting from the combination.

Type 2 diabetes remains the sixth leading cause of death in the US. Despite evolving technology and development of new medications, epidemiological data shows that only 37% of patients are in good glycemic control as defined by the American Diabetes Association. Recent large trials (UKPDS) suggest that any improvement in blood sugar control leads to favorable outcomes.

Human research suggests chromium improves insulin receptor sensitivity leading to blood sugar reduction. Research also shows blood levels of chromium are lower in people with type 2 diabetes and diabetic patients lose more chromium in their urine than people without diabetes.

This pilot trial will recruit type 2 diabetic subjects already on metformin and treat them with chromium picolinate for 8 weeks. The results of the trial will provide vital preliminary data including safety and size of effect to direct future, larger studies.

ELIGIBILITY:
Inclusion Criteria:

ICD-9 Diagnosis of TYpe 2 Diabetes (250.XX) for two years or less and treated with metformin Patients having completed dose titration of metformin as prescribed by their physician and have reached a stble dose between 1000-2550 mg per day for at least two months HbA1c: 7.0-10.5%

Exclusion Criteria:

* Duration of metformin treatment longer than 1 year at start time of study medication Historical or current use of oral anti-diabetes (OAD) medication (other than metformin) or use of insulin History ofmyocardial infarction within the lat 6 months, unstable angina, uncontrollable hypertension with systolic greater than 180 or diastolic greater than 110.

Clinical or objective finding suggestive of congestive heart failure. Individuals not receiving routine management by their primary car eproviders and/or endocrinologists for their type 2 diabetes, including routine ECG and ophthamological evaluations.

Women of child-bearing age not using standard birth control measures. Hemoglobin <11 or > 16; Hematocrig <32 or > 50; WBC <3,000 or >12,000; Platelets <150,000 or >500,000 Serum Creatinine >1.4 mg/dL; BUN >25 mg/dL Presence of greater than +1 protein on random macroscopic urinalysis at screening without a rule out of microalbuminuria Total bilirubin >1.5 mg/dL LFTs: AST>60 IU/L; ALT>65/L; Alkaline phosphatase >120 Iu/L. Isolated LFT elevations with an ultrasound diagnosis of non-alcoholic Steatohepatitis and a lab rule out of viral hepatitis will be included in the study with careful monitoring of LFTs.

Subjects currently taking nutritional supplements, including multivatmin for study duration; subjects will be asked to discontinue any nutritional supplementation at the screening telephone interview 1 week prior to screening lab work and 4 week sprior to baseline lab work.

Subjects taking lipid lowering medications except statins (i.e. niacin, fibrates, resins) due to possible chromium binding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-01; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Safety/Adverse Events
Hemoglobin A1c

SECONDARY OUTCOMES:
Fasting Blood Glucose, Fasting Insulin, HOMA Index
Lipid Profile: total cholesterol, LDL, HDL, Triglycerides
Oral Glucose Tolerance Test

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Bradley, ND, Principal Investigator — Bastyr University
Locations (2):
- United States (2):
  - Bastyr University Campus SPR, Kenmore, Washington
  - Bastyr Center for Natural Health, Seattle, Washington